CLINICAL TRIAL: NCT05931757
Title: A Multicenter, Prospective Clinical Study of Olverembatinib Combined With Blinatumomab in the Treatment of Adult de Novo Philadelphia Chromosome Positive Acute Lymphoid Leukemia
Brief Title: A Study of Olverembatinib Combined With Blinatumomab in the Treatment of Ph+ ALL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Principal Investigator, Chen Suning, Principal Investigator, The First Affiliated Hospital of Soochow University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ-ALL03
Record Dates: First submitted 2023-06-16; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Philadelphia-Positive ALL
MeSH Terms: interventions — olverembatinib; blinatumomab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment Group (Experimental): The patients would be treated with Olverembatinib, Given PO, combined with Blinatumomab, Given intravenously
  Interventions: Drug: Olverembatinib

INTERVENTIONS:
Drug: Olverembatinib — Olverembatinib will be taken 40mg qod from the time of diagnosis, and Blinatumomab will be given intravenously up to five cycles.
  Other Names: Blinatumomab

SUMMARY:
This is a multicenter, prospective, phase II study for adult de novo Philadelphia chromosome-positive acute lymphoid leukemia (Ph+ ALL) based on the combination of Olverembatinib and Blinatumomab. Olverembatinib will be taken 40mg qod from the time of diagnosis, and Blinatumomab will be given intravenously up to five cycles.

DETAILED DESCRIPTION:
This is a prospective, multicenter, one-arm phase II clinical study, aimed for evaluating the effectiveness and safety of Olverembatinib combined with Blinatumomab in the treatment of newly diagnosed adult Ph + ALL patients.

Subjects enrolled in this study will be given a 14-day induction regimen of Olverembatinib 40mg qod orally combined with blinatumomab. To prevent cytokine release syndrome (CRS), the subjects are permitted to receive pretreatment with dexamethasone combined with Olverembatinib until the leukocyte count is less than 5 × 109/L. During induction therapy, Blinatumomab will be given in an incremental dose regimen, i.e., 9 μ g/day on days 1 to 3 and 28 μ g/day was used on days 4 to 14, and then stopped for 14 days.

Olverembatinib 40mg qod combined with blinatumomab will subsequently administered as a consolidation regimen. Blinatumomab was given a fixed dose regimen during consolidation treatment, i.e. 28 μ g/day from the day 1 to the day 28, and then stopped for 14 days. A total of 3-4 cycles will be administered, with every 42 days as one cycle.

At the end of the consolidation treatment, the patient received a maintenance regimen of Olverembatinib 40mg qod orally for at least 5 years. If the patient loses molecular response (defined as BCR-ABL1/ABL1 > 0.10%) during maintenance treatment, another consolidation treatment of 3-4 cycles of blinatumomab will be initiated.

During induction and consolidation treatment, lumbar puncture combined with sheath injection will be performed three times every cycle to prevent central nervous system leukemia (CSNL). If CNSL occurs at the time of admission, patients should receive regular conventional lumbar puncture and sheath injection for treating CNSL.

During the treatment, each subject will be evaluated regularly, including hematological response, minimal residual disease (through flow cytology, FCM-MRD), cytogenetic response and molecular remission rate, as well as adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female patients who are 18 years of age or older.
2. Newly diagnosed Philadelphia chromosome-positive (Ph+) or BCR-ABL1-positive ALL, as defined by the 2016-WHO criteria. Participants should not be treated with any kind of TKIs or chemotherapy. Participants who only received preconditioning can be enrolled.
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2, and expected survival period ≥ 3 months.
4. Organ function as indicated by the following laboratory indicators must be met:

1) Alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN), aspartate aminotransferase (AST) ≤ 2.5 × ULN; 2) Total bilirubin≤1.5×ULN; 3) Serum creatinine≤1.5×ULN or 24-hour calculated creatinine clearance≥50mL/min when serum creatinine >1.5×ULN; 4) Amylase≤1.5×ULN, lipase≤1.5×ULN; 5) Cardiac ejection fraction (EF) > 50%, pulmonary artery systolic blood pressure ≤ 50mmHg; 6) QT interval corrected on electrocardiogram (ECG) evaluation: QTc≤450ms in males or ≤470ms in females; 7) PT, APTT and INR≤1.5×ULN.

5. Willingness and ability to comply with study procedures and follow-up examination.

Exclusion Criteria:

1. Human immunodeficiency virus (HIV) infection, or chronic infection with hepatitis B virus (HBsAg positive) or hepatitis C virus (anti-HCVpositive).
2. Uncontrolled active infection.
3. Patients who are currently suffering from active autoimmune disease or a history of autoimmune disease potentially involving the CNS.
4. Patients who have any history of heart or vascular disease, such as hypertension (systolic blood pressure(HBP) > 140mmHg and/or diastolic blood pressure > 90mmHg), or take medications that are known to cause QT interval prolongation. The patients with well controlled HBP can be considered to be included.
5. Cardiac ultrasonography indicates that pulmonary artery systolic blood pressure is >50 mmHg; or there are clinical symptoms related to pulmonary arterial hypertension.
6. Patients who suffer from severe bleeding disorders unrelated to Ph+ ALL.
7. Patients who have any other malignant tumors that require treatment.
8. Patients who have a history of pancreatitis or a history of alcohol abuse.
9. Patients who have severe hypertriglyceridemia (triglyceride ≥ 5.6mmol/L).
10. Patients who are pregnant, planning to become pregnant or breastfeeding.
11. Patients who underwent major surgery (except for minor surgery such as catheter placement or bone marrow biopsy) within 14 days before the first drug.
12. Patients who may not be able to complete all study visits or procedures required by the study protocol, including follow-up visits, and/or fail to comply with all required study procedures.
13. Patients who suffer from any condition or illness that, in the opinion of the Investigator, would compromise patient safety or interfere with the evaluation of the safety of the research drug.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Complete Molecular Remission. | From Induction through the end of three cycles of blinatumomab (approximately 16 weeks)
  Will be estimated along with the 95% credible intervals.

SECONDARY OUTCOMES:
Percentage of Participants with CR and Incomplete Complete Remission (CRi). | From Induction through the end of three cycles of blinatumomab (approximately 16 weeks)
  Will be estimated along with the 95% credible intervals.
Duration of Complete Molecular Remission. | From the date of acquisition of complete molecular remission until the date of loss of complete molecular remission, assessed up to 2 to 7 years.
  Will be estimated along with the 95% credible intervals.
Event-free survival (EFS) | From the first day of treatment until any failure (resistant disease, relapse, or death), assessed up to 2 to 7 years
  The Kaplan-Meier method will be used to assess EFS probabilities.
Overall survival (OS) | From the first day of treatment to time of death from any cause, assessed up 2 to 7 years.
  The Kaplan-Meier method will be used to assess OS probabilities.
Incidence of adverse events (AEs) | Up to approximately 2 to 7 years
  Will be graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. The proportion of patients with AEs will be estimated, along with the Bayesian 95% credible interval.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China